CLINICAL TRIAL: NCT00726310
Title: A Multicenter Prospective Patient Outcome Evaluation Of Spinelink® Fixation In The Treatment Of Degenerative Spondylolisthesis And Spinal Instability
Brief Title: Evaluation Of Spinelink® Fixation In The Treatment Of Degenerative Spondylolisthesis And Spinal Instability
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-044
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis
Keywords: Spondylolisthesis; Instability
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SpineLink® , SpineLink® II Group: Spinal fusion surgery with SpineLink®
  Interventions: Device: SpineLink® , SpineLink® II

INTERVENTIONS:
Device: SpineLink® , SpineLink® II — Spine plate system for lumbar spinal fusions

SUMMARY:
The purpose of this open, multi-center study is to prospectively collect outcome data on patients who are having lumbar spinal fusion surgery with implantation of the SpineLink® system.

DETAILED DESCRIPTION:
This will be an open, prospective, multi-center outcome study. This study will be conducted at up to ten centers, each of which will enroll approximately 20 patients. A maximum of 200 patients will be enrolled. This patient sample size will allow statistical comparison to historical literature and allow an inter-center comparison of outcome. Enrollment into the study may include all patients who have lumbar spinal fusion performed. All spinal fusion surgery will be performed using the EBI SpineLink® system.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has demonstrated Grade I or Grade II degenerative spondylolisthesis exhibited by maximum slippage on flexion and extension radiographs with symptoms that include back pain and/or leg pain with spinal fusion indicated, or spinal instability as evidenced by greater than 3 mm of translational motion or greater than 10 degrees of angular motion between the involved vertebrae as evidenced by flexion-extension radiographs.
2. This surgery will be the primary fusion attempt with no more than three (3) vertebrae or 2 disc spaces involved.
3. The patient must be available for yearly follow-up in the study until completion of the 24 month evaluation.
4. The patient must be skeletally mature (epiphyses closed).
5. Bone grafting material must be limited to autograft and/or bone-bank allograft.
6. The patient must be willing to comply with the treatment regimen, follow-up requirements, and have the legal ability to give informed consent.

Exclusion Criteria:

1. Patients with supplemental spinal internal fixation devices previously implanted at any other level and/or a previous fusion attempt at the involved level(s) (no interbody fusions, salvage procedures, or prior hardware).
2. Patients with other pathology at the involved spinal level, e.g., osteomyelitis, Paget's disease, pathologic fracture, etc.
3. Patients with a disease entity or condition that totally precludes the possibility of bony fusion such as known active cancer, etc.
4. Patients who have significant metabolic diseases including insulin dependent diabetes, renal dysfunction, etc.
5. Patients involved in personal injury litigation.
6. Pregnant or nursing females.
7. Patient in whom unapproved biologicals (e.g. BMP-2) or bone substitute materials (e.g. Grafton) would be used at the fusion site.
8. Patients who are unable to understand and sign an informed consent or who, in the opinion of the investigator, would be psychologically unwilling or unable to understand or complete the protocol, especially those unwilling or unable to participate in the follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Multiple site around the US
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2000-05; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Percentage of successful fusions achieved | 24 Months
  AP radiographs will be evaluated for the evidence of bridging virgin trabecular bone across the fusion mass. In order for a patient to be considered fused, A/P radiographs must show evidence of bridging virgin trabecular bone across the fusion mass.

SECONDARY OUTCOMES:
Neurologic Assessment | 24 Months
  Maintenance or Improvement
Radiographic Fusion Grade | 24 Months
  Radiographic fusion grade will be assessed at each follow up, as defined by Dawson et al. 8, as follows: A0 = Pseudarthrosis A1 = Unilateral Pseudarthrosis A2 = Insufficient Unilateral Bone Mass A3 = Contiguous Fusion without Hypertrophy A4 = Solid Fusion with Hypertrophy of Fusion Mass
SF-36 Health Survey | 24 Months
  Health Survey

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Alvarado Orthopedic Clinic, San Diego, California
  - Rogozinski Orthopedic Clinic, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: Undecided